CLINICAL TRIAL: NCT04112784
Title: Desaturation Validation of INVSENSOR00039
Status: Completed | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-20068
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- INVSENSOR00039 (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00039 sensor.
  Interventions: Device: INVSENSOR00039

INTERVENTIONS:
Device: INVSENSOR00039 — Noninvasive pulse oximeter sensor

SUMMARY:
This study is designed to compare the accuracy of a noninvasive measurement of oxygen saturation compared to reference values obtained by a laboratory blood gas analyzer. Arterial blood samples will be collected from healthy adult subjects while undergoing a desaturation procedure wherein the concentration of oxygen inhaled is slowly reduced. The subject will then be returned to breathing room air.

ELIGIBILITY:
Inclusion Criteria

* Subject is 18-50 years of age.
* Subject weighs a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
* Hemoglobin value is greater than or equal to 11 g/dL.
* Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
* Carbon monoxide (CO value) ≤ 2.0% fraction of carboxyhemoglobin (FCOHb)
* Subject has a physical status of ASA I or II (American Society of Anesthesiology Class I; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease) as it applies to the systemic disease portion of the classification.
* Blood pressure: Systolic Blood Pressure ≤ 140 mmHg and ≥ 90 mmHg, Diastolic Blood Pressure ≤ 90 mmHg and ≥ 50 mmHg, and if blood pressure is lower than 100/60 subject passes an orthostatic blood pressure test.
* Subject is able to read and communicate in English and understands the study and risks involved.

Exclusion Criteria (* = per physician discretion)

* Subject is pregnant.
* Subject has a Body Mass Index (BMI) > 35 and has been classified as morbidly obese or at an increased risk for participation by a medical professional.
* Subject has a history of fainting (vasovagal), blacking out or losing consciousness during or after blood draw, or has a fear of blood draws.
* Subject smokes one pack of cigarettes or more in one week, and/or the equivalent of e- cigarette liquid, and smokers are not being recruited as indicated in the Case Study Report Form (CSRF).
* Subject has open wounds, inflamed tattoos or piercings, and/or any visible healing wounds that a medical professional renders them at an increased risk for participation.*
* Subject has known drug or alcohol abuse and/or use of recreational drugs.
* Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
* Subject has experienced a concussion or head injury with loss of consciousness within the last 12 months.
* Subject has any history of a stroke, myocardial infarction, seizures or heart attack.
* Subject has a chronic bleeding disorder (i.e. hemophilia).
* Subject who has taken anticoagulant medication within the last 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDS)).
* Subject has donated blood within the past 4 weeks.
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
* Subject has any symptomatic cardiac dysrhythmia (i.e. atrial fibrillation) and has not received clearance by their physician to participate.
* Subject has a known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder, Multiple Sclerosis, Huntington's Disease) that interferes with the subject's level of consciousness.
* Subject has taken opioid pain medication 24 hours before the study.
* Subject has any type of infectious disease (i.e. Hepatitis, HIV, Tuberculosis, Flu, Malaria, Measles, etc.).
* Subject is taking medications known to treat any type of infectious disease.*
* Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
* Subject has had invasive surgery within the past year- including but not limited to major dental surgery*, appendix*, plastic surgery*.
* Subject has had invasive surgery within the past year- including but not limited to gallbladder, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, major ears, nose, and throat (ENT) surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
* Subject has symptoms of congestion, head cold, flu or other illnesses.
* Subject experiences claustrophobia or has generalized anxiety disorder.
* Subject has been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the last 12 months.
* Subject has any cancer or history of cancer (not including skin cancer).*
* Subject has chronic unresolved asthma, lung disease (including chronic obstructive pulmonary disease (COPD)) or respiratory disease.
* Subject is allergic to lidocaine, latex, adhesives, or plastic.
* Subject has heart conditions, insulin-dependent Diabetes or uncontrolled hypertension.
* Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the last 6 months.
* Subject intends on participating in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle, tennis) or exercise (working out, riding a bike, riding a skate board etc.), or any activity that will put additional stress on the wrist within 24 hours following a study that involves an arterial line.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00039
Started | 38
Completed | 25
Not Completed | 13
Not completed — Did Not Proceed Due to Time Constraints | 9
Not completed — Screen Failures | 4

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00039
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 4
  Black/African American | 6
  Caucasian | 10
  Hispanic | 5

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation (SpO2) Accuracy of Sensor
Description: Performance of the sensors will be determined by comparing the noninvasive oxygen saturation measurement (SpO2) of the pulse oximeter sensors to the arterial oxygen saturation (SaO2) value obtained from a reference blood sample and calculating the Accuracy root square mean (ARMS) value.
Time Frame: 1-5 hours
Measure: Number; unit: percentage of oxygen saturation
Arm/Group | INVSENSOR00039
Number analyzed (Participants) | 25
percentage of oxygen saturation | 1.0

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Arm/Group | INVSENSOR00039
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT04112784/Prot_SAP_000.pdf